CLINICAL TRIAL: NCT02132416
Title: Prospective Controlled Study of Surgical Management of Unstable Thoracic Cage Injuries and Chest Wall Deformity in Trauma
Brief Title: Operative Treatment of Unstable Thoracic Cage Injuries and Chest Wall Deformity in Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Eva-Corina Caragounis, MD, Sahlgrenska University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ec761218; epn887-13 (Registry Identifier: Regional Ethical Board)
Record Dates: First submitted 2014-05-01; First posted 2014-05-07 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Trauma; Flail Chest; Rib Fractures; Surgery
Keywords: Prospective study; Surgical management; Unstable thoracic cage injuries; Trauma; Ventilator support
MeSH Terms: conditions — Wounds and Injuries; Flail Chest; Rib Fractures | interventions — Anti-Inflammatory Agents, Non-Steroidal; Diclofenac; Naproxen; Ibuprofen; Analgesics, Opioid; Tramadol; Oxycodone; Morphine; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical management (Active Comparator): Operative fixation of unstable thoracic cage injuries and chest wall deformity. Thoracic Epidural anaesthesia will be offered. Paracetamol, Opioids and NSAID will be used as pain medication.
  Interventions: Drug: NSAID; Drug: Opioids; Drug: Thoracic Epidural anaesthesia; Drug: Paracetamol; Procedure: Surgical management
- Conservative management (Active Comparator): Conservative management of unstable thoracic cage injuries and chest wall deformity. Thoracic epidural anaesthesia will be offered. Paracetamol, Opioids and NSAID will be used as pain medication.
  Interventions: Drug: NSAID; Drug: Opioids; Drug: Thoracic Epidural anaesthesia; Drug: Paracetamol

INTERVENTIONS:
Drug: NSAID — Will be used if tolerated.
  Other Names: Diclofenac; Naprosyn; Ibuprofen
Drug: Opioids — Initially intravenous administration and when tolerated oral slow-release pils will be used.
  Other Names: Tramadol; Oxycodone; Morphine
Drug: Thoracic Epidural anaesthesia — Given by specialists in anaesthesiology and intensive care.
  Other Names: Continous thoracic epidural anaesthesia will be offered.
Drug: Paracetamol — 1g QID will be given to all patients unless allergies.
  Other Names: Paracet; Alvedon; Panodil
Procedure: Surgical management — Fracture stabilization
  Other Names: Matrix Rib Fixation System (DePuy Synthes).
  Arms: Surgical management

SUMMARY:
The purpose of this prospective controlled study is to determine whether surgical management of unstable thoracic cage injuries and chest wall deformity in trauma reduces the need for and the time spent on ventilator compared to a group treated without operation.

DETAILED DESCRIPTION:
Patients meeting the inclusion criteria and giving their informed consent will be enrolled in this prospective controlled study. Included patients at Sahlgrenska University Hospital will undergo surgical stabilization of chest wall injuries and patients at Karolinska University Hospital will be managed conservatively. A total of 60 patients will be included in each group. 3D reconstructions of computed tomography images of the Thorax done at admission to the hospital will be used in order to evaluate injury according to Lung Injury Scale and Chest wall Injury Scale and for calculating radiological lung volumes and plan surgical procedure in the intervention group. Surgery will be performed as soon as possible after inclusion. MatrixRIB® (DePuy Synthes) Fixation system is used for stabilizing rib fractures with plates and angular locked screws. In cases where thoracotomy is done the patients will receive an anterior and posterior chest tube and wound drain with active suction. All patients, both in the intervention and in the control group will be offered thoracic epidural anaesthesia. Broad-spectrum intravenous antibiotic therapy is given as long as the patient has chest tubes. Thrombotic prophylaxis with LMWH is given until the patient is mobilized but for a minimum of 7 days. Patients will be followed-up 6 weeks, 6 months and 1 year post-operatively by surgeon and physiotherapist. A low-dosage computer tomography of the thorax will be done after 6 months in order to evaluate healing of the rib cage, possible non-union or dysfunction of osteosynthetic material and measure remaining lung volume. This examination will be compared to the initial computer tomography image done when the patient was admitted. At follow-ups complaints, possible late complications, usage of analgesia and return to work will be recorded. Evaluated instruments, EQ-5D-5L, VAS with Pain-O-Meter (POM) and Disability Rating Index (DRI) will be used to evaluate quality of life, pain and physical function. Range of motion in the thorax, thoracic spine and shoulders will be evaluated for every patient. Breathing movements will be measured by using a Respiratory movement measuring instrument (RMMI, ReMo Inc) and lung function tests will be performed in a standardized manner.

In order to enrich the material, hospital data from patients fulfilling the inclusion criteria but not included, at the two study locations, during the inclusion period (June 2014 - June 2017) will be analyzed. An additional Ethical approval has been granted.

ELIGIBILITY:
Inclusion Criteria:

* Trauma with segmental rib fractures on at least 3 adjacent ribs ( anatomical flail chest )
* Trauma with chest wall deformity

Exclusion Criteria:

* Concurrent spinal cord injuries with paralysis
* Severe head injury where normal level of consciousness is not resumed
* Severe neurological and musculoskeletal diseases that influence the function of the thoracic wall and lung volumes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Respiratory insufficiency | 1 year
  Need and length of ventilation therapy

SECONDARY OUTCOMES:
Hospital stay | 6 weeks
  Time spent in an intensive care unit and total length of hospital stay

OTHER OUTCOMES:
Disability Rating Index | 1 year
  Pain, function and mobility
Quality of Life; EQ5D5L and VAS | Time Frame
  EQ-5D-5L instrument has a subscale of; 1 (no problems), 2 (slight problems), 3 (moderate problems), 4 (severe problems) and 5 (extreme problems). The Visual Analogue scale is a self-rating scale from 0% (the worst Health you can imagine) to 100% (the best Health you can imagine).

CONTACTS AND LOCATIONS:
Overall Officials: Hans Granhed, MD PhD, Study Director — Sahlgrenska University Hospital; Eva-Corina Caragounis, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (2):
- Sweden (2):
  - Departement of Surgery, Sahlgrenska University Hospital, Gothenburg
  - Departement of Intensive Care, Karolinska University Hospital, Stockholm

REFERENCES:
- [Derived] Caragounis EC, Fagevik Olsen M, Sandstrom L, Rossi Norrlund R, Strommer L, Granhed H. A bi-institutional observational study comparing short-term and long-term outcome of operative and non-operative management of clinical and radiological flail chest injuries. Scand J Trauma Resusc Emerg Med. 2025 May 15;33(1):87. doi: 10.1186/s13049-025-01400-8. PMID 40375321